CLINICAL TRIAL: NCT07267637
Title: "Autogenous Tooth Bone Graft for Alveolar Socket Preservation: A CBCT-Based Clinical Trial With 6-Month Follow-Up"
Brief Title: Autogenous Tooth Bone Graft for Alveolar Socket Preservation
Acronym: ATBG
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haifaa Mohammed Al-hussini (Other)
Responsible Party: Sponsor-Investigator, Haifaa Mohammed Al-hussini, "Principal Investigator, Haifaa Al-Hussini, BDS, MSc Candidate, Sana'a University", Sana'a University
Organization: Sana'a University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SU-DENT-ATBG-2025-HH
Record Dates: First submitted 2025-11-23; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Alveolar Bone Grafting; Bone Regeneration Following Wisdom Teeth Extraction; Tooth Extraction Site Healing
Keywords: Autogenous Tooth Bone Graft; Socket Preservation; CBCT Imaging; Bone Density Measurement; Bone Regeneration in Dentistry

STUDY DESIGN:
Intervention Model Description: This is a single-arm, open-label clinical trial designed to evaluate the efficacy of autogenous tooth bone grafts for alveolar socket preservation following sugrical tooth extraction. The intervention involves the use of the patient's own extracted tooth to prepare the bone graft, which will be placed into the extraction socket. The primary objective is to assess changes in alveolar bone height, width, and density before extraction and after six months of intervention using Cone Beam Computed Tomography (CBCT). All participants will undergo the same procedure, and no control group will be included. The study aims to explore the feasibility and outcomes of using autogenous grafts in dental socket preservation procedures
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autogenous Tooth Bone Graft Intervention Group (Experimental): "In this arm of the study, participants will receive an autogenous tooth bone graft for alveolar socket preservation following surgical tooth extraction. The intervention involves the extraction of the patient's own tooth, which will be processed and used as a bone graft. This graft will be placed into the empty socket immediately after the extraction. The purpose of this intervention is to prevent bone resorption, promote natural healing, and support bone regeneration within the extraction site. CBCT scans will be performed before extraction to measure baseline bone dimensions and will be repeated 6 months post-intervention to assess the success of bone preservation in terms of height, width, and density."
  Interventions: Biological: "Autogenous Tooth Bone Graft"

INTERVENTIONS:
Biological: "Autogenous Tooth Bone Graft" — "The intervention involves the use of the patient's own extracted tooth to create a bone graft for alveolar socket preservation following surgical tooth extraction. The patient's tooth is carefully processed to remove caries, periodontal ligaments, pulp, and any restorative materials, leaving behind a complete tooth structure (enamel, dentin, and cementum). This tooth is then crushed, disinfected, and treated before being placed into the empty socket. This graft helps maintain the structure of the alveolar bone by promoting natural bone regeneration and preventing resorption. The bone graft will be monitored for its efficacy in preserving alveolar bone height, width, and density, assessed using Cone Beam Computed Tomography (CBCT)."

SUMMARY:
The purpose of this clinical experiment is to assess how well autogenous tooth bone grafting preserves the alveolar socket after surgical tooth extraction. Before being inserted into the socket, the graft is made from the patient's own extracted tooth and ground into a particle. Twenty Yemeni patients who needed their teeth extracted are included in the trial, and they will be followed up with clinical and radiographic procedures using cone-beam computed tomography (CBCT) for six months. The primary objective is to ascertain whether the autogenous dental bone graft can preserve the height, width, and density of alveolar bone, offering a secure, affordable, and biocompatible substitute for traditional grafting materials.

DETAILED DESCRIPTION:
This interventional clinical study investigates the role of autogenous tooth bone graft in alveolar socket preservation after surgical tooth extraction. The extracted tooth is cleaned, dried, processed into particulate graft material manually using bone crusher, and disinfect and treated using (NaOH) and (Na CL). The graft particles are immediately placed into the fresh extraction socket and sutured. Twenty Yemeni patients requiring impacted lower third molar and upper canine teeth surgical extractions will be included. The healing process will be evaluated both clinically and radiographically over a 6-month period. Cone-beam computed tomography (CBCT) scans will be used to assess bone density and alveolar ridge dimensions before extraction and at six months' post-intervention. The study aims to determine whether autogenous tooth bone grafts can effectively reduce post-extraction alveolar bone resorption and maintain ridge dimensions, supporting their potential use as an autologous, biocompatible, and economically feasible graft material for clinical socket preservation.

ELIGIBILITY:
Inclusion Criteria:

* - Absence of systemic diseases.
* Very good to accepted oral hygiene.
* Patients with impacted teeth requiring extraction.
* Patients between the ages of 16 and 50.
* No history of smoking.
* No history of any other drug use.
* Patients who were cooperative, motivated, to attend the follow-up and maintenance visits.

Exclusion Criteria:

* Systemic conditions or pharmacological therapies that could be an absolute contraindication for the intervention (such as un controlled diabetics, immunocompromised states, or treatment with oral or parenteral bisphosphonates).
* Poor oral hygiene.
* Acute exacerbation of chronic infection like pain or swelling.
* Pregnant women, children, elderly (>60 years), physically and mentally challenged, terminally and seriously ill.
* Hight Smoking tendency.
* Patients who refused to participate in the trial.
* Uncooperative Patients who won't be able to maintain the follow up visits

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-07-14 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
"Alveolar Bone Height, Width, and Density Preservation with Autogenous Tooth Bone Graft" | "Before extraction and 6 months post-intervention"
  This study aims to evaluate the effectiveness of autogenous tooth bone grafts in preserving alveolar bone following tooth extraction. The study will assess changes in alveolar bone height, width, and density using Cone Beam Computed Tomography (CBCT) at two time points: before extraction (baseline) and 6 months post-grafting.
  The outcome measures are:
  Alveolar Bone Height: Measured in millimeters using CBCT at baseline and 6 months.
  Alveolar Bone Width: Measured in millimeters using CBCT at baseline and 6 months.
  Alveolar Bone Density: Measured in Hounsfield units using CBCT at both time points.
  The intervention involves using the patient's own extracted tooth to create a bone graft placed into the socket, promoting healing and bone regeneration. This study will determine the effectiveness of autogenous tooth bone grafts in preventing bone resorption and preserving alveolar socket structure.

CONTACTS AND LOCATIONS:
Overall Officials: Haifaa Alhussini, BDS, MSc, Principal Investigator — Sana'a University Faculty of Dentistry
Locations (1):
- Sana'a University faculty of Dentisrty, Sanaa, Sanaa Governorate, Yemen

IPD SHARING:
Plan to Share IPD: Yes
"We will share anonymized individual participant data (IPD), including baseline characteristics, clinical assessments, and key outcome measures (alveolar bone height, width, and density) collected before and after the autogenous tooth bone graft intervention. Access to the data will be granted to qualified researchers who meet the criteria for data sharing and comply with the applicable data use agreement."
Supporting Information: Study Protocol, SAP, ICF
Time Frame: "IPD and supporting information will be made available starting 12 months after the completion of the study. The data will be accessible for a period of 5 years."
Access Criteria: "Access to IPD and supporting information will be granted to qualified researchers who submit a data request via the ClinicalTrials.gov platform. Researchers must meet the criteria outlined in the Data Use Agreement, which ensures that the data will be used responsibly and for research purposes only."
URL: https://clinicaltrials.gov/

REFERENCES:
- [Result] Valdec S, Pasic P, Soltermann A, Thoma D, Stadlinger B, Rucker M. Alveolar ridge preservation with autologous particulated dentin-a case series. Int J Implant Dent. 2017 Dec;3(1):12. doi: 10.1186/s40729-017-0071-9. Epub 2017 Mar 30. PMID 28361377
- [Result] Mahardawi B, Damrongsirirat N, Dhanesuan K, Subbalekha K, Mattheos N, Pimkhaokham A. Radiographic changes after alveolar ridge preservation using autogenous raw tooth particles versus xenograft: A prospective controlled clinical trial. Clin Oral Implants Res. 2024 Dec;35(12):1597-1606. doi: 10.1111/clr.14348. Epub 2024 Aug 12. PMID 39132806
- See also: This study compares the effectiveness of autogenous raw tooth particles versus xenografts in preserving alveolar bone after tooth extraction. It uses radiographic assessments to evaluate bone resorption and preservation over time. The research provides i — https://pubmed.ncbi.nlm.nih.gov/28361377/
- See also: "This study discusses the use of autologous particulated dentin as a bone substitute for alveolar ridge preservation. The method demonstrates the potential of autologous dentin for bone augmentation in implant therapy, providing a viable alternative to x — https://pubmed.ncbi.nlm.nih.gov/39132806/
- Available data/document: Clinical Study Report: https://doi.org/10.1111/clr.14 — https://pubmed.ncbi.nlm.nih.gov/39132806/ — This data includes radiographic changes from the clinical trial involving alveolar ridge preservation using autogenous tooth particles and xenograft materials.
- Available data/document: Clinical Study Report: https://doi.org/10.1186/s40729 — https://pubmed.ncbi.nlm.nih.gov/28361377/ — "This study explores the use of autologous particulated dentin as a novel approach for alveolar ridge preservation. The intervention involves the patient's own extracted tooth, which is processed into dentin particles and used as a bone graft material. The study demonstrates successful outcomes in terms of bone regeneration and subsequent implant placement, suggesting that autologous dentin may be a promising alternative to traditional grafting materials.